CLINICAL TRIAL: NCT00789308
Title: Open Randomized Mult-Center Study to Evaluate Safety and Efficacy of Low Molecular Weight Sulfated Dextran in Islet Transplantation (CIT-01)
Brief Title: Safety and Effectiveness of Low Molecular Weight Sulfated Dextran in Islet Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Clinical Islet Transplantation Consortium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAIT CIT-01; CIT-01 (Other: Clinical Islet Transplantation Consortium); 2008-001210-25 (EudraCT Number)
Record Dates: First submitted 2008-11-10; First posted 2008-11-11 (Estimated); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Diabetes Mellitus, Type I
Keywords: Insulin dependence
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Heparin; Mycophenolic Acid; Sirolimus; Tacrolimus; Cyclosporine; thymoglobulin; Antilymphocyte Serum; Basiliximab; Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of Care (Active Comparator): 18 participants randomized to protocol immunosuppression (Daclizumab OR Basiliximab; Tacrolimus OR Cyclosporine; Mycophenolate Mofetil OR Sirolimus; and heparin) without LMW-DS
  Interventions: Drug: Heparin; Drug: CellCept® (Mycophenolate mofetil) OR Rapamune® (Sirolimus); Drug: Prograf® (Tacrolimus) OR Cyclosporine; Drug: Thymoglobulin® (Anti-thymocyte Globulin) - at first transplant; Drug: Simulect® (Basiliximab) - at 2nd or 3rd transplant; Drug: Klexane® (Enoxaparinsodium); Drug: Trombyl® or Albyl-E® (Acetylsalicylicacid- ASA); Drug: Enbrel® (Etanercept)
- LMW-DS (Experimental): 18 participants randomized to protocol immunosuppression (Daclizumab OR Basiliximab; Tacrolimus OR Cyclosporine; Mycophenolate Mofetil OR Sirolimus; and heparin) and LMW-DS
  Interventions: Drug: Low Molecular Weight Sulfated Dextran (LMW-SD); Drug: CellCept® (Mycophenolate mofetil) OR Rapamune® (Sirolimus); Drug: Prograf® (Tacrolimus) OR Cyclosporine; Drug: Thymoglobulin® (Anti-thymocyte Globulin) - at first transplant; Drug: Simulect® (Basiliximab) - at 2nd or 3rd transplant; Drug: Klexane® (Enoxaparinsodium); Drug: Trombyl® or Albyl-E® (Acetylsalicylicacid- ASA); Drug: Enbrel® (Etanercept)

INTERVENTIONS:
Drug: Low Molecular Weight Sulfated Dextran (LMW-SD) — Inhibitor of IBMIR
  Arms: LMW-DS
Drug: Heparin — Anticoagulation
  Arms: Standard of Care
Drug: CellCept® (Mycophenolate mofetil) OR Rapamune® (Sirolimus) — Cell proliferation inhibitor
Drug: Prograf® (Tacrolimus) OR Cyclosporine — Calcineurin inhibitor
Drug: Thymoglobulin® (Anti-thymocyte Globulin) - at first transplant
Drug: Simulect® (Basiliximab) - at 2nd or 3rd transplant — Monoclonal IL-2 receptor blocker
Drug: Klexane® (Enoxaparinsodium) — Anticoagulation Prophylaxis
Drug: Trombyl® or Albyl-E® (Acetylsalicylicacid- ASA) — Anticoagulation Prophylaxis
Drug: Enbrel® (Etanercept) — Anti-Inflammatory Therapy

SUMMARY:
Type 1 diabetes is an autoimmune disease in which the insulin-producing pancreatic beta cells are destroyed, resulting in poor blood sugar control. The purpose of this study is to assess the safety and effectiveness of low molecular weight sulfated dextran (LMW-SD) on post-transplant islet function in people with type 1 diabetes who have responded to intensive insulin therapy.

DETAILED DESCRIPTION:
Type I diabetes, also known as insulin-dependent diabetes, is a chronic disease in which the pancreas produces insufficient insulin to properly regulate blood sugar levels. Hypoglycemia, or low blood sugar, and hyperglycemia, or high blood sugar, can lead to significant complications in people with type 1 diabetes. Intensive insulin therapy has been shown to reduce the risk of chronic complications in people who achieve near normalization of glycemia. However, this therapy is labor intensive, difficult to implement, and associated with an increased frequency of severe hypoglycemia. Transplantation of islets from a healthy pancreas has been successful in restoring normal blood sugar levels and has led to initial insulin independence in people with type 1 diabetes. Rejection of these islets by the recipient's immune system, however, can make the treatment ineffective. An immune response known as instant blood-mediated inflammatory reaction (IBMIR) results in the disruption of islet integrity and islet loss within an hour of transfusion. LMW-SD inhibits IBMIR by preventing the cascade that triggers it, when combined with pancreatic islets. The purpose of this study is to determine the safety and efficacy of LMW-SD given with islet transfusion and post-transfusion along with immunosuppressive therapy, including mycophenolate mofetil or sirolimus, tacrolimus or cyclosporine, and thymoglobulin or basiliximab, on the success of islet transplantation in people with type 1 diabetes.

This study will last for 1 year after the final islet transplant. Participants may receive up to 3 islet transplants while participating in this study. Participants eligible for this study will have clinic visits every 6 months. Once a preparation of islets becomes available, participants will be randomly assigned to Arm 1 or Arm 2. Participants in Arm 1 will receive LMW-DS during and for 5 hours after infusion. Participants in Arm 2 will receive heparin at the time of infusion. In addition, all participants will receive anticoagulation prophylaxis agents consisting of Klexzane® (Enoxaparinsodium) and Trombyl® or Albyl-E® (Acetylsalicylic acid). All participants will also receive the oral immunosuppression medications consisting of mycophenolate mofetil or sirolimus and tacrolimus or cyclosporine throughout the study. In addition, they will receive intravenous thymoglobulin on days -2, -1, day 0 (transplant), +1, and +2 for the first transplant or intravenous basiliximab at the time of transplant and on Day 4 for the second and third transplant. Enbrel® (Etanercept) will be given to all participants for anti-inflammatory therapy. Islet infusions will occur at the hospital and will be given intravenously. Participants will be eligible to receive second and third islet infusions if previous infusions fail and they continue to meet the eligibility criteria. After each infusion, study visits will occur on Days 1, 3, 7, 14, 21, 28, and 75 and Months 6 and 12. At these visits, physical exams and blood collection will occur. At some visits, urine collection will also occur.

ELIGIBILITY:
Inclusion Criteria:

* Mentally stable and able to comply with study procedures;
* Clinical history compatible with type 1 diabetes, with:

  * onset of disease at less than 40 years of age,
  * insulin dependence for at least 5 years at study entry, and
  * sum of age and insulin-dependent diabetes duration of at least 28.
* Absent stimulated C-peptide (less than 0.3 ng/ml) 60 and 90 minutes post-mixed-meal tolerance test;
* Involvement of intensive diabetes management, defined as:

  * Self-monitoring of glucose values no less than a mean of three times each day, averaged over each week,
  * Administration of three or more insulin injections each day or insulin pump therapy,
  * Under the direction of an endocrinologist, diabetologist, or diabetes specialist, with at least three clinical evaluations during the past 12 months.
* At least one episode of severe hypoglycemia in the past 12 months, defined as an event with symptoms compatible with hypoglycemia in which the individual required assistance of another person and which was associated with either a blood glucose level less than 54 mg/dl or prompt recovery after an oral carbohydrate, intravenous glucose, or glucagon administration; and
* Reduced awareness of hypoglycemia OR marked glycemic lability OR a composite of a Clarke score of 3 or more or a HYPO score greater or equal to the 75th percentile in the 12 months prior to randomization.

Exclusion Criteria:

* Known IgE mediated allergy to antibiotics used in the culture medium;
* Known hypersensitivity to dextran;
* Body mass index (BMI) greater than 30 kg/m^2;
* Insulin requirement of more than 1.0 IU/kg/day;
* HbA1c greater than 10%;
* Untreated proliferative diabetic retinopathy;
* Systolic blood pressure higher than 160 mmHg or diastolic blood pressure higher than 100 mmHg;
* Measured glomerular filtration rate (GFR) using 51Cr-EDTA, 99technetium-DPTA, or iohexol of less than 80 ml/min/1.73m^2;
* Presence or history of macroalbuminuria (greater than 300 mg/g creatinine);
* Presence or history of panel-reactive anti-HLA antibody levels greater than 20% by flow cytometry;
* Pregnant, breastfeeding, or unwilling to use effective contraception throughout the study and for 4 months after study completion;
* Active infection, including hepatitis B virus, hepatitis C virus, HIV, or tuberculosis;
* Negative for Epstein-Barr virus by IgG determination;
* History of malignancy with exception of completely resected squamous or basal cell carcinoma of the skin;
* Known active alcohol or substance abuse;
* Baseline Hgb below the lower limits of normal, lymphopenia, neutropenia, or thrombocytopenia;
* Activated protein C resistance (APC-R);
* Any coagulopathy or individuals with an INR greater than 1.5;
* Severe coexisting cardiac disease, characterized by any one of the following conditions:

  * Heart attack within the last 6 months,
  * Evidence of ischemia on functional heart exam within the year prior to study entry, or
  * Left ventricular ejection fraction less than 30%.
* Persistent elevation of liver function tests at the time of study entry;
* Acute or chronic pancreatitis;
* Active peptic ulcer disease, symptomatic gallstones, or a history of portal hypertension;
* Severe unremitting diarrhea, vomiting, or other gastrointestinal disorders that could interfere with the ability to absorb oral medications;
* Currently receiving treatment for a medical condition that requires chronic use of systemic steroids;
* Treatment with any antidiabetic medication other than insulin, within 4 weeks prior to study entry;
* Use of any investigational medications within the past 4 weeks;
* Received a live attenuated vaccine within the past 2 months;
* Treatment with any immunosuppressive regimen at time of study entry;
* Previous islet transplant;
* Previous pancreas transplant.

  --Note: Participants who had a pancreas transplant more than 6 months prior to study entry that failed within the first week due to thrombosis, followed by surgical removal of the transplanted pancreas, are not excluded.
* Or any medical condition that, in the opinion of the investigator, might interfere with safe participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-07-11 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2014-08-21 (Actual)

PRIMARY OUTCOMES:
Level of stimulated c-peptide at 90-minute derived from the mixed-meal tolerance test (MMTT) | At 70 to 80 days after first islet transfusion

SECONDARY OUTCOMES:
Number of participants who achieve and maintain a 7.0% HbA1c level | Throughout Study
Number of severe hypoglycemic events | Throughout study
Percent reduction in insulin requirements | At 70 to 80 days after first islet transfusion, At 365 days after first and final islet infusion
Ryan hypoglycemia severity score ( HYPO) score | : At 70 to 80 days after first islet transfusion, At 365 days after first and final islet infusion
Proportion of participants with full graft function | At 70 to 80 days after first islet transfusion and after the final islet infusion
C-peptide to glucose creatinine ratio | At 70 to 80 days after first islet transfusion, At 365 days after first and final islet infusion
Proportion of participants receiving a second islet infusion and proportion of participants receiving a third islet transfusion | At 70 to 80 days after first islet transfusion and after the final islet infusion
Incidence and severity of adverse events related to islet infusion procedure | At 70 to 80 days and 350 to 379 days after the first islet transfusion
Incidence of worsening retinopathy | At 350 to 379 days after the first islet transfusion
HbA1c level | At 70 to 80 days after first islet transfusion, At 365 days after first and final islet infusion
Mean amplitude of glycemic excursions (MAGE) | At 70 to 80 days after first islet transfusion, At 365 days after first and final islet infusion
Glycemic lability index (LI) | At 70 to 80 days after first islet transfusion, At 365 days after first and final islet infusion
Clarke hypoglycemia awareness score | At 70 to 80 days after first islet transfusion, At 365 days after first and final islet infusion
Basal (fasting) and 90-minute glucose and c-peptide derived from MMTT | : At 70 to 80 days after first islet transfusion, At 365 days after first and final islet infusion
Beta-score | At 70 to 80 days after first islet transfusion, At 365 days after first and final islet infusion
Acute insulin response to glucose, insulin sensitivity, and disposition index derived from the insulin-modified frequently-sampled intravenous glucose tolerance (FSIGT) test, | At 70 to 80 days after first islet transfusion, At 365 days after first and final islet infusion
Glucose variability and hypoglycemic duration derived from continuous glucose monitoring system(CGMS) | At 70 to 80 days after first islet transfusion, At 365 days after first and final islet infusion
Incidence of a change in the immunosuppression drug regimen | At 70 to 80 days and 350 to 379 days after the first islet transfusion
Incidence of immune sensitization defined by detecting anti-HLA antibodies not present prior to transplantation | At 70 to 80 days and 350 to 379 days after the first islet transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Olle Korsgren, MD, Principal Investigator — Uppsala University Hospital, Sweden; Torbjörn Lundgren, MD, Study Chair — Karolinska University Hospital
Locations (3):
- University Hospital Rikshospitalet, Oslo, Norway
- Sweden (2):
  - Karolinska University Hospital, Stockholm
  - Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share data upon completion of the study in: Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: On average, within 24 months after database lock for the trial.
Access Criteria: Open access.
URL: https://www.immport.org/home

REFERENCES:
- [Result] von Zur-Muhlen B, Lundgren T, Bayman L, Berne C, Bridges N, Eggerman T, Foss A, Goldstein J, Jenssen T, Jorns C, Morrison Y, Ryden M, Schwieger T, Tufveson G, Nilsson B, Korsgren O. Open Randomized Multicenter Study to Evaluate Safety and Efficacy of Low Molecular Weight Sulfated Dextran in Islet Transplantation. Transplantation. 2019 Mar;103(3):630-637. doi: 10.1097/TP.0000000000002425. PMID 30211831
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) — https://www.niddk.nih.gov/
- See also: Clinical Islet Transplantation Consortium website — https://www.citisletstudy.org/
- Available data/document: Individual Participant Data Set: Accession ID: SDY1437 — https://www.immport.org/shared/study/SDY1437 — Digital object identifier (DOI): 10.21430/M3YZY4PXCS. Location of data: Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.
- Available data/document: Study Protocol: Accession ID: SDY1437 — https://www.immport.org/shared/study/SDY1437 — Digital object identifier (DOI): 10.21430/M3YZY4PXCS. Location of data: Immunology Database and Analysis Portal (ImmPort).
- Available data/document: Statistical Analysis Plan: Accession ID: SDY1437 — https://www.immport.org/shared/study/SDY1437 — Digital object identifier (DOI): 10.21430/M3YZY4PXCS. Location of data: Immunology Database and Analysis Portal (ImmPort).
- Available data/document: Informed Consent Form: Accession ID: SDY1437 — https://www.immport.org/shared/study/SDY1437 — Digital object identifier (DOI): 10.21430/M3YZY4PXCS. Location of data: Immunology Database and Analysis Portal (ImmPort).